CLINICAL TRIAL: NCT05597462
Title: A Randomized, Double-blind Trial Evaluating the Effects of Treatment With DFD-29 Capsules 40 mg QD in Comparison to Placebo on Microbial Flora in Healthy Adult Human Subjects, When Administered Over a Period of 16 Weeks.
Brief Title: Impact of DFD-29 on Microbial Flora of Healthy, Adult Human Subjects When Administered Over 16 Weeks
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Journey Medical Corporation (Industry)
Collaborators: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: DFD-29-CD-006
Record Dates: First submitted 2022-10-24; First posted 2022-10-28 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-08

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea | interventions — Minocycline

STUDY DESIGN:
Intervention Model Description: A multi-center, randomized, double-blind, placebo-controlled, parallel group trial with a treatment period of 16 weeks.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DFD-29 (Experimental): DFD-29 (minocycline hydrochloride) capsules, 40 mg will be administered orally once daily for 16 weeks.
  Interventions: Drug: Minocycline hydrochloride capsules
- Placebo (Placebo Comparator): Placebo capsules will be administered orally once daily for 16 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Minocycline hydrochloride capsules — Minocycline hydrochloride capsules, 40 mg will be administered orally once daily for 16 weeks.
  Other Names: DFD-29
  Arms: DFD-29
Other: Placebo — Placebo capsules will be administered orally once daily for 16 weeks.
  Other Names: Placebo comparator
  Arms: Placebo

SUMMARY:
The purpose of this trial is to evaluate the effects of 16-week treatment with DFD-29 40 mg QD dose in comparison to Placebo on the skin, intestinal and vaginal microbiota.

DETAILED DESCRIPTION:
A multi-center (up to three sites), randomized, double-blind, placebo-controlled, parallel group trial with a treatment period of 16 weeks.

Sixty (60) healthy adult human subjects will be randomized in a 2:1 ratio to receive treatment with DFD-29 (Minocycline Hydrochloride Capsules) 40 mg QD orally or matching Placebo (for DFD-29 capsules) QD orally for a period of 16 weeks.

The trial will have a screening period (Day -30 to Day -1) and a trial treatment period (Day 1 to Day 113). There will be 6 planned visits to the study site for subjects.

Impact on microbial flora will be assessed from skin swabs, stool samples and vaginal swabs (female subjects) taken at multiple timepoints.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant, non-lactating female aged ≥ 18 and ≤ 65 years.
2. Subjects must have understood, and signed IRB/IEC approved written ICF.
3. Subjects must be willing to refrain from using all other antibiotics during the 16-week treatment period, other than the IP.
4. Women of childbearing potential* must not be pregnant or lactating at the time of screening visit as documented by a negative urine pregnancy test.
5. Women of childbearing potential must be willing to use an acceptable form of birth control during the trial from the day of the first dose administration to 30 days after the last administration of trial drug.
6. All male subjects must agree to use accepted methods of birth control with their partners, throughout the study and until 30 days after the last administration of trial drug.
7. Subjects must be in good health and free from any clinically significant disease, which may interfere with the evaluation of microbiota or the administration of the IP.

Exclusion Criteria:

1. Female subjects who are pregnant, lactating or planning to become pregnant during trial participation.
2. History of allergy or known sensitivity to minocycline, doxycycline, other tetracycline, or any component of the study medication.
3. Clinically significant abnormal laboratory test results that, in the opinion of the Investigator, would compromise the subject's safety or ability to participate in the trial
4. History of organ transplant requiring immunosuppression, HIV, or other immune compromised state.
5. History of lupus-like syndrome, autoimmune hepatitis, vasculitis, or serum sickness.
6. Any clinically significant condition that, in the opinion of the Investigator, would interfere with the study evaluations or would place the trial subject at undue safety risk.
7. Subjects with an active acute or chronic systemic infections
8. Subjects with planned surgery during the trial or within 30 days after the last dose administration
9. Subjects who cannot avoid excessive exposure to UV radiation (use of tanning booths or extended /occupational exposure to sunlight)
10. Subjects that have a medical history of photosensitivity or hyperpigmentation
11. Female subjects with medical history within 3 months prior to randomization of having vaginitis or that use a vaginal douche or vaginal cleaning agent within 48 hours of any visit
12. Subjects who used the following

    1. Non-tetracycline antibiotics (systemic) within 6 weeks prior to Baseline (BL)
    2. Tetracycline antibiotics (systemic) within 3 months prior to BL
13. Subjects who consume excessive amounts of alcohol (greater than two drinks per day) or use drugs of abuse (including, but not limited to, cannabinoids, cocaine and barbiturates) within one year prior to screening
14. Subjects who have been treated with systemic retinoids or therapeutic Vitamin A supplements > 10,000 IU/ day (multivitamin tablets are allowed) within 180 days prior to the BL
15. Subjects who are on anti-coagulants or those likely to require anti-coagulants during the trial period
16. Subjects who have used methoxyflurane or other nephrotoxic drugs (in the opinion of the Investigator) within the past 30 days of BL
17. Subjects who have used topical retinoids or topical antibiotics to the face 30 days prior to BL
18. Subjects who have used on their facial skin within 30 days prior to BL topical corticosteroids, topical anti-mycotic, topical azelaic acid or ivermectin
19. Subjects who have participated in an investigational drug trial (i.e., subjects have been treated with an investigational drug) within 30 days prior to BL or where sufficient washout period has not been achieved; whichever period is longer.
20. Subjects having symptoms of COVID-19 or have had close contact with someone with suspected or confirmed SARS-CoV-2 infection within 10 days prior to screening or who are at high risk of SARS-CoV-2 infection.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Changes in the number of colony forming units (CFUs) of microbial species. | Baseline to Week 16
  Change in the colony forming units (CFUs) of microbial species colonized from skin, gastrointestinal or vaginal swabs from Baseline (BL) to Week 16 in comparison of DFD-29 versus Placebo treatment groups
Changes in MIC90 of selected colonized microbial species. | Baseline to Week 16.
  Changes in MIC90 of the selected colonized microbial species to minocycline in the comparison of DFD-29 group versus Placebo treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Srinivas Sidgiddi, M.D., Study Director — Journey Medical Corporation
Locations (2):
- United States (2):
  - 3A Research, LLC, Las Cruces, New Mexico
  - 3A Research, LLC, El Paso, Texas

IPD SHARING:
Plan to Share IPD: Yes
We will comply with the HIPAA regulations in this matter.
Supporting Information: Study Protocol, SAP
Time Frame: Before database lock for the study